CLINICAL TRIAL: NCT04996836
Title: Evaluating the Predictive and Prognostic Power of the Early Breast canceR gEnetic and Epigenetic Abnormalities Through Liquid biopSy and neTwOrk MEdicine Algorithm: the BR(E)2ASTOME Phase II Randomized Controlled Trial
Brief Title: Breast Cancer, Omics, and Precision Medicine
Acronym: BR(E)2ASTOME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Giuditta Benincasa, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: LV
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Liquid biopsy; DNA methylation; Omics; Biomarkers; Network Analysis; Precision Medicine
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BC diagnosis and Omics (Experimental): Participants will be offered:
  1. Liquid biopsy of ctDNA and targeted NGS (BRCA1, BRCA2, CHEK2, PALB2, BRIP1, TP53, PTEN, STK11, CDH1, ATM, BARD1, MLH1, MRE11A, MSH2, MSH6, MUTYH, NBN, PMS1, PMS2, RAD50, RAD51C, RAD51D, NF1, EPCAM, SMARCA4, CDK12);
  2. Whole-genome RRBS
  Interventions: Biological: Next Generation Sequencing and Network Analysis
- BC diagnosis and standard of the care (No Intervention): Participants will not be offered targeted NGS or whole-genome RRBS but will receive their usual clinical care

INTERVENTIONS:
Biological: Next Generation Sequencing and Network Analysis — Next Generation Sequencing and Network Analysis will profile genetic and epigenetic abnormalities in blood from patients with BC.
  Arms: BC diagnosis and Omics

SUMMARY:
The standard tissue biopsy strategy for cancer detection is not comprehensive enough to profile the whole epi-genomic signatures of breast cancer (BC) and ensure an accurate prognosis and prediction of drug response. Liquid-based assays have the potential to reduce the molecular heterogeneity of BC and a possible utility for improving disease management. In particular, genomic DNA (gDNA) and circulating tumor (ctDNA) can be sequenced for genetic and epigenetic (DNA methylation) profiling of the BC patients to enhance personalized prognosis and prediction of drug therapy. We describe a study protocol for evaluating the clinical utility of the early use of the network-oriented BR(E)2ASTOME algorithm which combine the power of liquid-based assays, advanced epi-genomics platform, and network analysis to identify improve precision medicine and personalized therapy of BC.

DETAILED DESCRIPTION:
The BR(E)2ASTOME study will be performed at the U.O.C. Patologia Molecolare e Clinica, University of Campania "L. Vanvitelli", Naples (Italy) with a long-standing experience in diagnosis and treatment of BC (Refs.). From each study participant, total of 10 mL of pheripheral blood in EDTA tubes will be collected at time of BC diagnosis. Blood-based assays will be performed to obtain genetic and/or epigenetic big data from ct-DNA and gDNA, respectively. A network-oriented algorithm combined with patient-level clinical information will be applied to big data in order to identify clusters of genes (BC-modules) harboring novel genetic mutations, in the NGS-ctDNA BC-group, and differentially methylated regions (DMRs), in the RRBS-gDNA group, with a potential predictive and prognostic role in BC management. In the NGS-ctDNA-RRBS-gDNA group, we will evaluate whether the multi-omics approach is more informative as compared to the single-omic paradigm.

BC patients (males and females) will be randomized to the 2 study arms: ctDNA-NGS + gDNA-RRBS, and standard of care alone. No modifications of intervention assignment will be possible after randomization process of patients. The BR(E)2ASTOME study will provide evidence about the potential clinical utility of early use liquid-based assays and network-oriented biomarkers in prognosis and prediction of drug response in BC management.

Thus, results from BR(E)2ASTOME study will bring to identify not only new molecular mechanisms associated with BC, but also non-invasive biomarkers that can direct towards an early diagnosis, contribute to monitor the cancer progression and the response to therapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sporadic BC
* Inherited BC
* 18 years old
* Males and Females

Exclusion Criteria:

* Inflammatory diseases
* Cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Network-oriented buomarkers in prognosis of BC | 1 years
  We will evaluate whether the network-oriented BR(E)2ASTOME approach will identify BC modules useful for a better stratification of BC severity.
  We will measure:
  DNA methylation levels and associations with clinical parameters (survival, hospitalization, all-cause mortality).
  We will evaluate potential novel genetic mutations in targeted genes and associations with clinical parameters (survival, rate of hospitalization, all-cause mortality)
Evaluation of Network-oriented buomarkers of Drug Response | 2 years
  We will evaluate whether the network-oriented BR(E)2ASTOME approach will identify BC modules useful for predicting the individual drug response.
  We will measure DNA methylation levels, and potential novel genetic mutations, and their association with clinical parameters (poor/good response to drug therapy).

IPD SHARING:
Plan to Share IPD: No